CLINICAL TRIAL: NCT04690075
Title: Dietary Fiber in Nutritional Therapy for Chronic Diseases
Brief Title: Effect of Dietary Fiber on Metabolism, Inflammation and Nutritional Status in Patients With Chronic Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Yu Kang, MD, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DFiber-CD-2020-2021
Record Dates: First submitted 2020-12-14; First posted 2020-12-30 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Chronic Disease; Dietary Fiber
Keywords: dietary fiber; chronic disease; metabolism; inflammation; nutritional status
MeSH Terms: conditions — Chronic Disease; Inflammation | interventions — Nutrition Therapy; Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): To receive routine nutrition management and dietary fiber supplements based on recommendation for 12 weeks.
  Interventions: Dietary Supplement: Nutrition Management and Dietary Fiber
- Control (Placebo Comparator): To receive routine nutrition management for 12 weeks.
  Interventions: Dietary Supplement: Nutrition Management

INTERVENTIONS:
Dietary Supplement: Nutrition Management and Dietary Fiber — Routine nutrition management and dietary fiber supplements based on recommendation for 12 weeks.
  Arms: Intervention
Dietary Supplement: Nutrition Management — Routine nutrition management for 12 weeks.
  Arms: Control

SUMMARY:
The prevalence of chronic disease is increasing rapidly in China. Medical nutritional therapy (MNT) is essential for the prevention and control of chronic diseases. For example, dietary fiber plays an important role in chronic disease management. Evidence suggests that increasing fiber intake can decrease the risk of chronic diseases, such as overweight/obesity, hyperlipidemia, hyperglycemia, GI diseases, etc. However, according to the nation-wide survey, the dietary fiber intake of Chinese people shows a downward trend in recent years, and the relationship between dietary fiber and metabolism of chronic patients is still controversial. So, this study aims to explore the effects of dietary fiber on metabolism, inflammatory factors and nutritional status among patients with chronic diseases, so as to provide reference for proper nutrition intervention towards chronic disease.

DETAILED DESCRIPTION:
Investigators plan to recruit potential participants in hospital clinics using posters. An anticipated total of 120 patients with chronic diseases (including overweight, obesity, hyperlipemia, hyperglycemia, etc) will be randomized to receive oat beta-glucans (study group) or routine nutrition management (control group) respectively. The outcome parameters, including weight, blood glucose level, blood fat level, etc, will be measured and compared over a 12-week intervention period. Intention-to-treat analysis (ITT) and per-protocol analysis (PP) will be conducted in statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70y
* Be diagnosed with obesity, hyperlipemia or hyperglycemia
* Fully understood and voluntarily signed the informed consent

Exclusion Criteria:

* Secondary hyperlipidemia or hyperglycemia
* Multiple organ failure
* Allergic or intolerant to dietary fiber(dietary supplement)
* Have gastrointestinal diseases
* Have a history of abdominal diseases
* Experienced intra-abdominal surgery
* Pregnant and lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-12-24 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of total cholesterol (TC) level | baseline, 12 weeks
  Total cholesterol (TC) level obtained from laboratory test
Change of low density lipoprotein (LDL) cholesterol level | baseline, 12 weeks
  Low density lipoprotein (LDL) cholesterol level obtained from laboratory test

SECONDARY OUTCOMES:
Change of interleukin-6 (IL-6) level | baseline, 12 weeks
  Interleukin-6 (IL-6) level obtained from laboratory test
Change of tumor necrosis factor-alpha level | baseline, 12 weeks
  Change of tumor necrosis factor-alpha level obtained from laboratory test
Change of triglyceride (TG) level | baseline, 12 weeks
  Change of triglyceride (TG) level obtained from laboratory test
Change of high density lipoprotein (HDL) cholesterol level | baseline, 12 weeks
  Change of high density lipoprotein (HDL) cholesterol level obtained from laboratory test
Change of fasting blood glucose (FBG) level | baseline, 12 weeks
  Change of fasting blood glucose (FBG) level obtained from laboratory test
Change of 2 hours postprandial blood glucose level | baseline, 12 weeks
  Change of 2 hours postprandial blood glucose level obtained from laboratory test
Change of hemoglobin level | baseline, 12 weeks
  Change of hemoglobin level obtained from laboratory test
Change of total body fat level | baseline, 12 weeks
  Change of total body fat level obtained from bioelectrical impedance analysis
Change of Percent of body fat (PBF) level | baseline, 12 weeks
  Change of percent of body fat (PBF) level obtained from bioelectrical impedance analysis
Change of visceral fat area (VFA) level | baseline, 12 weeks
  Change of visceral fat area (VFA) level obtained from bioelectrical impedance analysis

CONTACTS AND LOCATIONS:
Overall Officials: Kang Yu, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang L, Gao P, Zhang M, Huang Z, Zhang D, Deng Q, Li Y, Zhao Z, Qin X, Jin D, Zhou M, Tang X, Hu Y, Wang L. Prevalence and Ethnic Pattern of Diabetes and Prediabetes in China in 2013. JAMA. 2017 Jun 27;317(24):2515-2523. doi: 10.1001/jama.2017.7596. PMID 28655017
- [Background] Baigent C, Keech A, Kearney PM, Blackwell L, Buck G, Pollicino C, Kirby A, Sourjina T, Peto R, Collins R, Simes R; Cholesterol Treatment Trialists' (CTT) Collaborators. Efficacy and safety of cholesterol-lowering treatment: prospective meta-analysis of data from 90,056 participants in 14 randomised trials of statins. Lancet. 2005 Oct 8;366(9493):1267-78. doi: 10.1016/S0140-6736(05)67394-1. Epub 2005 Sep 27. PMID 16214597
- [Background] Ren J, Grundy SM, Liu J, Wang W, Wang M, Sun J, Liu J, Li Y, Wu Z, Zhao D. Long-term coronary heart disease risk associated with very-low-density lipoprotein cholesterol in Chinese: the results of a 15-Year Chinese Multi-Provincial Cohort Study (CMCS). Atherosclerosis. 2010 Jul;211(1):327-32. doi: 10.1016/j.atherosclerosis.2010.02.020. Epub 2010 Feb 21. PMID 20223457
- [Background] Pop-Busui R, Boulton AJ, Feldman EL, Bril V, Freeman R, Malik RA, Sosenko JM, Ziegler D. Diabetic Neuropathy: A Position Statement by the American Diabetes Association. Diabetes Care. 2017 Jan;40(1):136-154. doi: 10.2337/dc16-2042. No abstract available. PMID 27999003
- [Background] Nutrition recommendations and principles for people with diabetes mellitus. American Diabetes Association. J Fla Med Assoc. 1998 Aug;85(2):25-9. PMID 9782716
- [Background] Holman RR, Paul SK, Bethel MA, Matthews DR, Neil HA. 10-year follow-up of intensive glucose control in type 2 diabetes. N Engl J Med. 2008 Oct 9;359(15):1577-89. doi: 10.1056/NEJMoa0806470. Epub 2008 Sep 10. PMID 18784090